CLINICAL TRIAL: NCT05493111
Title: A Long-Term Safety Study Evaluating the Safety and Systemic Exposure of AR-15512, a Cold Thermoreceptor Modulator, for the Treatment of Dry Eye Disease (COMET-4)
Brief Title: A Long-Term Safety Study Evaluating the Safety and Systemic Exposure of AR-15512
Acronym: COMET-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-15512-LTSS
Record Dates: First submitted 2022-07-26; First posted 2022-08-09 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.003% AR-15512 (Experimental): 0.003% AR-15512 ophthalmic solution, one drop in each eye twice a day for 365 days
  Interventions: Drug: 0.003% AR-15512 ophthalmic solution
- AR-15512 Vehicle (Placebo Comparator): AR-15512 vehicle ophthalmic solution, one drop in each eye twice a day for 365 days
  Interventions: Drug: AR-15512 vehicle ophthalmic solution

INTERVENTIONS:
Drug: 0.003% AR-15512 ophthalmic solution — Active ingredients administered via topical ocular instillation
  Arms: 0.003% AR-15512
Drug: AR-15512 vehicle ophthalmic solution — Inactive ingredients administered via topical ocular instillation
  Arms: AR-15512 Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety of topical ophthalmic 0.003% AR-15512 compared to its vehicle dosed twice daily (BID) in subjects with dry eye disease (DED) for 12 months.

DETAILED DESCRIPTION:
At the end of the Screening Visit, subjects will undergo a protocol-specified washout period for prohibited prior and concomitant therapies. At the Baseline Visit, subjects who qualify based on inclusion/exclusion criteria will be enrolled in the study and randomized in a 2:1 ratio to receive 0.003% AR-15512 or AR-15512 Vehicle administered as 1 drop in each eye twice a day for 365 days (12 months). At the end of the Day 365 visit, subjects will exit the study.

Aerie Pharmaceuticals was acquired by Alcon on November 22, 2022.

ELIGIBILITY:
Key Inclusion Criteria:

* Previous history of Dry Eye Disease (DED) within the previous 12 months of the Baseline visit.
* Have used or desired to use artificial tears for DED symptoms within 3 months prior to the Baseline visit.
* Corrected visual acuity as specified in the protocol at the Baseline visit.
* Good general and ocular health, as determined by the investigator using medical history, ophthalmic examination and history, and vital signs (heart rate and blood pressure) at the Baseline visit.

Key Exclusion Criteria:

* History or presence of any ocular disorder or condition (other than DED) in either eye that would, in the opinion of the investigator, likely interfere with the interpretation of the study results or subject safety.
* Current evidence of other significant ophthalmic disease requiring topical medication (e.g. glaucoma, ocular hypertension) which may interfere with vision (e.g., cataract, macular degeneration) or other disease which the investigator believes may interfere with study findings or interpretation.
* Use of contact lenses in either eye within 7 days prior to the Baseline visit or planned use during the study.
* Use of medications as specified in the protocol.
* Use of lid heating therapy (i.e., LipiFlow®, iLUX®) or Meibomian gland probing/therapeutic expression within 6 months prior to the Baseline visit or anticipated during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scientific Advisor, CRD, Study Director — Alcon Research, LLC
Locations (10):
- United States (10):
  - Arizona Eye Center, Chandler, Arizona
  - Arizona Eye Institute, Sun City, Arizona
  - Global Research Management, Glendale, California
  - Macy Eye Center, Los Angeles, California
  - Eye Research Foundation, Newport Beach, California
  - Shultz Vision, Northridge, California
  - SightMD, Manhasset, New York
  - University Eye Specialists, Maryville, Tennessee
  - Piedmont Eye Center, Lynchburg, Virginia
  - Periman Eye Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 10 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all subjects who signed an informed consent and met all eligibility criteria.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Started | 182; 364 eyes | 93; 186 eyes
Completed | 149; 298 eyes | 76; 152 eyes
Not Completed | 33; 66 eyes | 17; 34 eyes
Not completed — Adverse Event | 3 | 4
Not completed — Withdrawal of Consent | 19 | 10
Not completed — Non-compliance | 1 | 1
Not completed — Lost to Follow-up | 8 | 1
Not completed — Disallowed Concurrent Treatment | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All randomized subjects who have received at least one dose of the study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle | Total
Number analyzed (Participants) | 182 | 93 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (14.46) | 59.1 (15.42) | 60.5 (14.79)
Age, Customized [Number; unit: subjects]
  18-29 years | 5 | 4 | 9
  30 to 45 years | 23 | 16 | 39
  46-60 years | 44 | 23 | 67
  61-75 years | 81 | 42 | 123
  Greater than 75 years | 29 | 8 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 65 | 195
  Male | 52 | 28 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 21 | 58
  Not Hispanic or Latino | 145 | 72 | 217
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: subjects]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 16 | 10 | 26
  Black or African American | 23 | 14 | 37
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 138 | 67 | 205
  Multi-racial | 0 | 0 | 0
  Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Ocular Treatment-Emergent Adverse Events by Preferred Term With Incidence Greater Than 2 Percent
Description: A treatment-emergent adverse event was defined as any event that occurred or worsened on or after the day randomized study intervention was initiated. At each study visit, subjects were verbally asked by clinic staff to report any changes to any aspect of their ocular health. Ocular treatment-emergent adverse events reported by the subject or observed by the investigator were summarized by preferred term for overall incidence calculation. This was a subject-based assessment.
Time Frame: Day 1 post-treatment, up to Day 365
Population: Safety Population
Measure: Number; unit: adverse event
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 182 | 93
adverse event
  Instillation site pain | 90 | 7
  Eye pruritis | 2 | 3
  Eyelid margin crusting | 1 | 2

2. Primary Outcome: Mean Change From Baseline in Heart Rate at Each Study Visit
Description: Heart rate was measured using manual or automated methods and recorded in beats per minute (bpm). Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 175 | 88
beats per minute
  Change from Baseline at Day 14 | 0.7 (9.06) | 0.6 (8.51)
  Change from Baseline at Day 90: number analyzed (Participants) | 169 | 84
  Change from Baseline at Day 90 | 1.4 (9.04) | 1.7 (10.93)
  Change from Baseline at Day 180: number analyzed (Participants) | 153 | 76
  Change from Baseline at Day 180 | 0.5 (9.20) | -0.9 (9.71)
  Change from Baseline at Day 270: number analyzed (Participants) | 148 | 74
  Change from Baseline at Day 270 | 0.8 (9.57) | 0.5 (9.34)
  Change from Baseline at Day 365: number analyzed (Participants) | 148 | 76
  Change from Baseline at Day 365 | 1.1 (9.73) | 1.0 (10.00)

3. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure at Each Study Visit
Description: Systolic blood pressure was measured using an appropriate sphygmomanometer and recorded in millimeters mercury (mmHg). Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 175 | 88
mmHg
  Change from Baseline at Day 14 | 1.4 (16.62) | 1.7 (14.40)
  Change from Baseline at Day 90: number analyzed (Participants) | 169 | 84
  Change from Baseline at Day 90 | 0.0 (14.27) | 1.2 (14.65)
  Change from Baseline at Day 180: number analyzed (Participants) | 153 | 76
  Change from Baseline at Day 180 | -3.3 (15.23) | 0.1 (17.19)
  Change from Baseline at Day 270: number analyzed (Participants) | 148 | 74
  Change from Baseline at Day 270 | -1.3 (14.98) | -1.8 (16.38)
  Change from Baseline at Day 365: number analyzed (Participants) | 148 | 76
  Change from Baseline at Day 365 | 0.1 (16.25) | -0.3 (13.65)

4. Primary Outcome: Mean Change From Baseline in Diastolic Blood Pressure at Each Study Visit
Description: Diastolic blood pressure was measured using an appropriate sphygmomanometer and recorded in millimeters mercury (mmHg). Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 175 | 88
mmHg
  Change from Baseline at Day 14 | 1.7 (9.29) | 0.6 (9.81)
  Change from Baseline at Day 90: number analyzed (Participants) | 169 | 84
  Change from Baseline at Day 90 | 0.2 (9.73) | 1.1 (9.63)
  Change from Baseline at Day 180: number analyzed (Participants) | 153 | 76
  Change from Baseline at Day 180 | 1.1 (9.01) | 1.6 (9.96)
  Change from Baseline at Day 270: number analyzed (Participants) | 148 | 74
  Change from Baseline at Day 270 | 0.8 (9.63) | 0.5 (9.83)
  Change from Baseline at Day 365: number analyzed (Participants) | 148 | 76
  Change from Baseline at Day 365 | 1.4 (9.56) | 1.3 (9.23)

5. Primary Outcome: Mean Change From Baseline in Overall Average Endothelial Cell Density at Day 365
Description: Cell density in the central corneal endothelium was assessed using specular microscopy imaging. Overall average cell density was calculated as the average of the average cell densities of three images and was measured in cells per millimeter squared (cells/mm^2). A negative change from baseline represents a less desirable outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: cells/mm^2
Units Other Than Participants: eyes
Groups:
- 0.003% AR-15512 - Right Eye; 0.003% AR-15512 - Left Eye: 0.003% AR-15512 ophthalmic solution, one drop in each eye twice a day for 365 days
- AR-15512 Vehicle - Right Eye; AR-15512 Vehicle - Left Eye: AR-15512 vehicle ophthalmic solution, one drop in each eye twice a day for 365 days
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 145 | 146 | 76 | 76
Number analyzed (eyes) | 145 | 146 | 76 | 76
cells/mm^2 | 12.8 (204.06) | 32.4 (203.12) | -40.4 (172.29) | -15.7 (162.02)

6. Primary Outcome: Percentage of Subjects With 10 Percent or More Decrease From Baseline in Overall Average Endothelial Cell Density at Study Exit
Description: Cell density in the central corneal endothelium was assessed using specular microscopy imaging. Overall average cell density was calculated as the average of the average cell densities of three images and was measured in cells per millimeter squared (cells/mm^2). A decrease from baseline represents a less desirable outcome.
Time Frame: Baseline (Day 1 pretreatment), Study Exit (Day 365, early termination visit, or unscheduled visit)
Population: Safety Population with data at baseline and corresponding visit
Measure: Number; unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 151 | 152 | 79 | 79
Number analyzed (eyes) | 151 | 152 | 79 | 79
percentage of subjects | 3.3 | 2.6 | 5.1 | 2.5

7. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Basophil Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Basophil level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9 cells/L)
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
10^9 cells per liter (10^9 cells/L)
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | 0.00 (0.057) | -0.01 (0.052)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -0.01 (0.053) | -0.01 (0.048)

8. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Basophils to Leukocytes Ratio Reported in Percentage of Cells
Description: A small volume of blood was collected and sent to a laboratory for analysis. The basophils to leukocytes ratio was reported as the absolute number of basophils divided by the absolute number of leukocytes multiplied by 100. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
percentage of cells
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | 0.03 (0.256) | 0.02 (0.291)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -0.05 (0.217) | -0.02 (0.238)

9. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Eosinophil Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Eosinophil level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
10^9 cells/L
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | 0.02 (0.143) | 0.01 (0.084)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | 0.02 (0.150) | 0.00 (0.076)

10. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Eosinophils to Leukocytes Ratio Reported in Percentage of Cells
Description: A small volume of blood was collected and sent to a laboratory for analysis. The eosinophils to leukocytes ratio was reported as the absolute number of eosinophils divided by the absolute number of leukocytes multiplied by 100. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
percentage of cells
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | 0.29 (1.626) | 0.20 (1.468)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | 0.34 (2.081) | 0.13 (1.333)

11. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Erythrocyte Mean Corpuscular Hemoglobin Concentration Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Erythrocyte mean corpuscular hemoglobin concentration level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 136 | 64
grams per liter (g/L)
  Change from Baseline at Day 180: number analyzed (Participants) | 136 | 62
  Change from Baseline at Day 180 | -2.0 (9.45) | -1.3 (8.71)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | 1.2 (8.76) | 0.9 (9.74)

12. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Erythrocyte Mean Corpuscular Hemoglobin Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Erythrocyte mean corpuscular hemoglobin level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 136 | 64
picograms (pg)
  Change from Baseline at Day 180: number analyzed (Participants) | 136 | 62
  Change from Baseline at Day 180 | -0.01 (1.020) | 0.01 (0.609)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | 0.21 (0.877) | 0.26 (0.905)

13. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Erythrocyte Mean Corpuscular Volume
Description: A small volume of blood was collected and sent to a laboratory for analysis. Erythrocyte mean corpuscular volume was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: femtoliters (fL)
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 136 | 64
femtoliters (fL)
  Change from Baseline at Day 180: number analyzed (Participants) | 136 | 62
  Change from Baseline at Day 180 | 0.53 (2.996) | 0.33 (2.548)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | 0.28 (2.449) | 0.50 (2.684)

14. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Erythrocyte Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Erythrocyte level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12 cells/L)
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 136 | 64
10^12 cells per liter (10^12 cells/L)
  Change from Baseline at Day 180: number analyzed (Participants) | 136 | 62
  Change from Baseline at Day 180 | -0.071 (0.2858) | -0.036 (0.2738)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -0.073 (0.2873) | -0.076 (0.2347)

15. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Erythrocyte Distribution Width Reported as Percentage of Variation of Cells
Description: A small volume of blood was collected and sent to a laboratory for analysis. Erythrocyte distribution width was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: percentage of variation of cells
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 136 | 64
percentage of variation of cells
  Change from Baseline at Day 180: number analyzed (Participants) | 136 | 62
  Change from Baseline at Day 180 | 0.09 (1.038) | 0.13 (0.721)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -0.02 (0.924) | -0.17 (0.666)

16. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Hematocrit Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Hematocrit level was reported as the volume of red blood cells in liters (L) divided by the volume of blood in L. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: proportion
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 136 | 64
proportion
  Change from Baseline at Day 180: number analyzed (Participants) | 136 | 62
  Change from Baseline at Day 180 | -0.0038 (0.02449) | -0.0020 (0.02580)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -0.0053 (0.02723) | -0.0051 (0.02443)

17. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Hemoglobin Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Hemoglobin level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 136 | 64
g/L
  Change from Baseline at Day 180: number analyzed (Participants) | 136 | 62
  Change from Baseline at Day 180 | -2.1 (7.94) | -1.1 (8.38)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -1.3 (8.69) | -1.3 (7.91)

18. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Leukocyte Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Leukocyte level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 136 | 64
10^9 cells/L
  Change from Baseline at Day 180: number analyzed (Participants) | 136 | 62
  Change from Baseline at Day 180 | -0.06 (1.653) | -0.46 (1.054)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -0.12 (1.351) | -0.38 (1.342)

19. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Lymphocyte Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Lymphocyte level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
10^9 cells/L
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | -0.28 (0.500) | -0.28 (0.522)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -0.18 (0.417) | -0.32 (0.466)

20. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Lymphocytes to Leukocytes Ratio Reported in Percentage of Cells
Description: A small volume of blood was collected and sent to a laboratory for analysis. The lymphocytes to leukocytes ratio was reported as the absolute number of lymphocytes divided by the absolute number of leukocytes multiplied by 100. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
percentage of cells
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | -3.21 (6.934) | -1.76 (6.713)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -1.95 (6.664) | -2.20 (6.544)

21. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Monocyte Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Monocyte level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
10^9 cells/L
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | -0.02 (0.148) | -0.03 (0.145)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -0.01 (0.167) | -0.01 (0.185)

22. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Monocytes to Leukocytes Ratio Reported in Percentage of Cells
Description: A small volume of blood was collected and sent to a laboratory for analysis. The monocytes to leukocytes ratio was reported as the absolute number of monocytes divided by the absolute number of leukocytes multiplied by 100. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
percentage of cells
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | -0.10 (2.100) | 0.21 (2.005)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | 0.09 (2.182) | 0.25 (2.040)

23. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Neutrophil Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Neutrophil level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
10^9 cells/L
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | 0.20 (1.532) | -0.17 (0.912)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | 0.05 (1.208) | -0.05 (1.197)

24. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Neutrophils to Leukocytes Ratio Reported in Percentage of Cells
Description: A small volume of blood was collected and sent to a laboratory for analysis. The neutrophils to leukocytes ratio was reported as the absolute number of neutrophils divided by the absolute number of leukocytes multiplied by 100. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
percentage of cells
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | 3.00 (8.231) | 1.32 (8.546)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | 1.58 (8.055) | 1.84 (7.839)

25. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Platelet Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Platelet level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 63
10^9 cells/L
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | -3.9 (42.18) | -9.0 (40.42)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 63
  Change from Baseline at Day 365 | -3.7 (32.58) | -1.5 (39.96)

26. Primary Outcome: Mean Change From Baseline in Hematology by Visit - Mean Platelet Volume
Description: A small volume of blood was collected and sent to a laboratory for analysis. Platelet volume was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 135 | 64
fL
  Change from Baseline at Day 180: number analyzed (Participants) | 135 | 62
  Change from Baseline at Day 180 | -0.24 (0.511) | -0.15 (0.559)
  Change from Baseline at Day 365: number analyzed (Participants) | 125 | 64
  Change from Baseline at Day 365 | -0.04 (0.479) | -0.24 (0.433)

27. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Alanine Aminotransferase Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Alanine aminotransferase level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 145 | 71
units per liter (U/L)
  Change from Baseline at Day 180 | 0.3 (15.01) | -2.5 (12.11)
  Change from Baseline at Day 365: number analyzed (Participants) | 141 | 71
  Change from Baseline at Day 365 | -0.2 (13.38) | -1.4 (12.59)

28. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Albumin Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Albumin level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 148 | 73
g/L
  Change from Baseline at Day 180 | -2.0 (2.37) | -1.9 (2.56)
  Change from Baseline at Day 365: number analyzed (Participants) | 143 | 73
  Change from Baseline at Day 365 | -2.1 (2.35) | -2.1 (2.30)

29. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Alkaline Phosphatase Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Alkaline phosphatase level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 148 | 73
U/L
  Change from Baseline at Day 180 | 2.5 (13.12) | 0.4 (16.66)
  Change from Baseline at Day 365: number analyzed (Participants) | 143 | 73
  Change from Baseline at Day 365 | -1.3 (16.12) | -3.5 (13.59)

30. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Aspartate Aminotransferase Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Aspartate aminotransferase level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 145 | 71
U/L
  Change from Baseline at Day 180 | 0.6 (14.74) | -0.1 (7.80)
  Change from Baseline at Day 365: number analyzed (Participants) | 141 | 71
  Change from Baseline at Day 365 | 0.0 (11.98) | 0.1 (9.39)

31. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Calcium Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Calcium level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 148 | 73
millimoles per liter (mmol/L)
  Change from Baseline at Day 180 | -0.044 (0.1051) | -0.037 (0.1026)
  Change from Baseline at Day 365: number analyzed (Participants) | 143 | 73
  Change from Baseline at Day 365 | -0.049 (0.1114) | -0.055 (0.0923)

32. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Creatinine Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Creatinine level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: micromoles per liter (Umol/L)
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 148 | 73
micromoles per liter (Umol/L)
  Change from Baseline at Day 180 | 1.3 (13.69) | -0.2 (12.38)
  Change from Baseline at Day 365: number analyzed (Participants) | 143 | 73
  Change from Baseline at Day 365 | 6.0 (60.26) | 1.3 (10.00)

33. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Globulin Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Globulin level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 148 | 73
g/L
  Change from Baseline at Day 180 | 0.3 (2.61) | 0.5 (2.44)
  Change from Baseline at Day 365: number analyzed (Participants) | 143 | 73
  Change from Baseline at Day 365 | 0.0 (2.43) | -0.1 (2.05)

34. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Potassium Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Potassium level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 133 | 69
mmol/L
  Change from Baseline at Day 180: number analyzed (Participants) | 133 | 66
  Change from Baseline at Day 180 | 0.09 (0.492) | 0.11 (0.482)
  Change from Baseline at Day 365: number analyzed (Participants) | 132 | 69
  Change from Baseline at Day 365 | 0.06 (0.470) | 0.16 (0.704)

35. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Protein Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Protein level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 148 | 73
g/L
  Change from Baseline at Day 180 | -1.7 (4.19) | -1.4 (4.15)
  Change from Baseline at Day 365: number analyzed (Participants) | 143 | 73
  Change from Baseline at Day 365 | -2.1 (3.97) | -2.2 (3.67)

36. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Sodium Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Sodium level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 148 | 73
mmol/L
  Change from Baseline at Day 180 | 0.0 (2.46) | -0.1 (2.17)
  Change from Baseline at Day 365: number analyzed (Participants) | 143 | 73
  Change from Baseline at Day 365 | 0.4 (2.36) | 0.5 (2.11)

37. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Triglyceride Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Triglyceride level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 148 | 73
mmol/L
  Change from Baseline at Day 180 | 0.079 (1.1354) | -0.276 (1.1943)
  Change from Baseline at Day 365: number analyzed (Participants) | 143 | 73
  Change from Baseline at Day 365 | -0.024 (0.9164) | -0.120 (1.2344)

38. Primary Outcome: Mean Change From Baseline in Chemistry by Visit - Urea Nitrogen Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Urea nitrogen level was measured. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 148 | 72
mmol/L
  Change from Baseline at Day 180 | 0.22 (2.066) | 0.06 (1.889)
  Change from Baseline at Day 365: number analyzed (Participants) | 143 | 72
  Change from Baseline at Day 365 | 0.16 (2.372) | 0.044 (1.637)

39. Primary Outcome: Mean Change From Baseline in Urinalysis by Visit - Specific Gravity Level
Description: A small volume of blood was collected and sent to a laboratory for analysis. Specific gravity level was calculated by dividing the sample's density by the density of water. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 140 | 66
ratio
  Change from Baseline at Day 180: number analyzed (Participants) | 140 | 65
  Change from Baseline at Day 180 | 0.0005 (0.00783) | 0.0020 (0.00713)
  Change from Baseline at Day 365: number analyzed (Participants) | 130 | 66
  Change from Baseline at Day 365 | 0.0007 (0.00886) | 0.0019 (0.00732)

40. Primary Outcome: Mean Change From Baseline in Urinalysis by Visit - pH Level
Description: A small volume of urine was collected and sent to a laboratory for analysis. The pH scale ranges from 0 (most acidic) to 14 (most alkaline), with 7 as neutral. Minimal change from the start of the study indicates a better outcome.
Time Frame: Baseline (Day 1 pretreatment), Day 180, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | 0.003% AR-15512 | AR-15512 Vehicle
Number analyzed (Participants) | 140 | 66
pH
  Change from Baseline at Day 180: number analyzed (Participants) | 140 | 65
  Change from Baseline at Day 180 | 0.06 (0.882) | -0.02 (0.857)
  Change from Baseline at Day 365: number analyzed (Participants) | 130 | 66
  Change from Baseline at Day 365 | 0.05 (0.712) | 0.03 (0.769)

41. Primary Outcome: Mean Best Corrected Visual Acuity (BCVA) Letter Score by Visit
Description: Visual acuity with correction in place (spectacles or a trial frame with lenses) was measured using Early Treatment Diabetic Retinopathy Study (ETDRS) letter charts (original or modified) at a distance of 10 feet. Each line on the ETDRS chart typically has five letters, and each letter correctly identified adds to the overall score. ETDRS letter scores range from 0 to 100, with each letter correctly identified representing a score of 1. A perfect score of 100 is achieved when all 70 letters on the chart are correctly identified. 85 letters correctly identified corresponds to normal distance eyesight.
Time Frame: Baseline (Day 1 pretreatment), Day 365
Population: Safety Population with data at visit
Measure: Mean (Standard Deviation); unit: letter
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 181 | 181 | 93 | 93
Number analyzed (eyes) | 181 | 181 | 93 | 93
letter
  Baseline | 84.9 (5.38) | 84.7 (6.05) | 85.8 (5.19) | 84.9 (5.91)
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eyes) | 149 | 149 | 76 | 76
  Day 365 | 85.1 (6.23) | 84.6 (7.15) | 84.9 (5.89) | 84.1 (5.90)

42. Primary Outcome: Mean Corrected Visual Acuity in LogMar by Visit
Description: Visual acuity with correction in place (spectacles or a trial frame with lenses) was measured using Early Treatment Diabetic Retinopathy Study (ETDRS) letter charts (original or modified) at a distance of 10 feet. Each line on the ETDRS chart typically has five letters, and each letter correctly identified adds to the overall score. The overall letter score was converted to Logarithmic minimum angle of resolution (LogMAR). LogMAR scores typically range from -0.3 to 1.0, where zero represents normal vision, negative values indicate better than normal vision, and positive values indicate poorer than normal vision.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eyes) | 182 | 182 | 93 | 93
logMAR
  Baseline | 0.062 (0.1326) | 0.061 (0.1339) | 0.064 (0.1433) | 0.080 (0.1435)
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eyes) | 175 | 175 | 88 | 88
  Day 14 | 0.055 (0.1386) | 0.053 (0.1406) | 0.048 (0.1334) | 0.053 (0.1481)
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eyes) | 169 | 169 | 84 | 84
  Day 90 | 0.046 (0.1315) | 0.044 (0.1279) | 0.048 (0.1339) | 0.049 (0.1268)
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eyes) | 153 | 153 | 76 | 76
  Day 180 | 0.047 (0.1304) | 0.045 (0.1298) | 0.042 (0.1523) | 0.051 (0.1548)
  Day 270: number analyzed (Participants) | 147 | 147 | 74 | 74
  Day 270: number analyzed (eyes) | 147 | 147 | 74 | 74
  Day 270 | 0.076 (0.1364) | 0.070 (0.1288) | 0.065 (0.1461) | 0.092 (0.1458)
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eyes) | 149 | 149 | 76 | 76
  Day 365 | 0.063 (0.1183) | 0.060 (0.1244) | 0.080 (0.1523) | 0.084 (0.1460)

43. Primary Outcome: Number of Subjects With Clinically Significant Biomicroscopy Findings as Determined by the Investigator at Each Study Visit - Lid Erythema
Description: An eye exam (slit lamp biomicroscopy) was performed by the investigator at each study visit. Findings related to lid erythema (redness of the eyelid) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
subjects
  Baseline | 1 | 1 | 0 | 0
  88Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  88Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  88Day 14 | 0 | 0 | 0 | 1
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Day 90 | 0 | 0 | 0 | 0
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Day 180 | 0 | 0 | 0 | 0
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 0 | 0 | 0 | 1
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 0 | 0 | 0 | 0

44. Primary Outcome: Number of Subjects With Clinically Significant Biomicroscopy Findings as Determined by the Investigator at Each Study Visit - Lid Edema
Description: An eye exam (slit lamp biomicroscopy) was performed by the investigator at each study visit. Findings related to lid edema (swelling of the eyelid) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
subjects
  Baseline | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  Day 14 | 0 | 0 | 0 | 0
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Day 90 | 1 | 1 | 0 | 0
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Day 180 | 0 | 0 | 0 | 0
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 0 | 0 | 0 | 0
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 0 | 0 | 0 | 0

45. Primary Outcome: Number of Subjects With Clinically Significant Biomicroscopy Findings as Determined by the Investigator at Each Study Visit - Conjunctiva Hyperemia
Description: An eye exam (slit lamp biomicroscopy) was performed by the investigator at each study visit. Findings related to conjunctiva hyperemia (increased amount of blood in the conjunctiva) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
subjects
  Baseline | 2 | 2 | 0 | 0
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  Day 14 | 0 | 0 | 0 | 0
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Day 90 | 1 | 1 | 0 | 0
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Day 180 | 0 | 0 | 1 | 0
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 1 | 0 | 0 | 0
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 0 | 0 | 0 | 0

46. Primary Outcome: Number of Subjects With Clinically Significant Biomicroscopy Findings as Determined by the Investigator at Each Study Visit - Conjunctiva Edema
Description: An eye exam (slit lamp biomicroscopy) was performed by the investigator at each study visit. Findings related to conjunctiva edema (swelling of the conjunctiva) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
subjects
  Baseline | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  Day 14 | 0 | 0 | 0 | 0
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Day 90 | 0 | 0 | 0 | 0
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Day 180 | 0 | 0 | 0 | 0
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 0 | 0 | 0 | 0
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 0 | 0 | 0 | 0

47. Primary Outcome: Number of Subjects With Clinically Significant Biomicroscopy Findings as Determined by the Investigator at Each Study Visit - Cornea Staining/Erosion
Description: An eye exam (slit lamp biomicroscopy) was performed by the investigator at each study visit. Findings related to cornea staining/erosion were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
subjects
  Baseline | 2 | 2 | 0 | 0
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  Day 14 | 0 | 0 | 0 | 0
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Day 90 | 0 | 0 | 0 | 0
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Day 180 | 0 | 0 | 0 | 0
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 0 | 0 | 0 | 0
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 0 | 0 | 0 | 0

48. Primary Outcome: Number of Subjects With Clinically Significant Biomicroscopy Findings as Determined by the Investigator at Each Study Visit - Cornea Edema
Description: An eye exam (slit lamp biomicroscopy) was performed by the investigator at each study visit. Findings related to cornea edema (swelling of the cornea) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
subjects
  Baseline | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  Day 14 | 0 | 0 | 0 | 0
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Day 90 | 0 | 0 | 0 | 0
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Day 180 | 0 | 0 | 0 | 0
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 0 | 0 | 0 | 0
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 0 | 0 | 0 | 0

49. Primary Outcome: Number of Subjects With Clinically Significant Biomicroscopy Findings as Determined by the Investigator at Each Study Visit - Anterior Chamber Cells
Description: An eye exam (slit lamp biomicroscopy) was performed by the investigator at each study visit. Findings related to cells in the anterior chamber (the fluid-filled space located in the front of the eye between the cornea and the iris) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
subjects
  Baseline | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  Day 14 | 0 | 0 | 0 | 0
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Day 90 | 0 | 0 | 0 | 0
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Day 180 | 0 | 0 | 0 | 0
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 0 | 0 | 0 | 0
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 0 | 0 | 0 | 0

50. Primary Outcome: Number of Subjects With Clinically Significant Biomicroscopy Findings as Determined by the Investigator at Each Study Visit - Anterior Chamber Flare
Description: An eye exam (slit lamp biomicroscopy) was performed by the investigator at each study visit. Findings related to anterior chamber flare (a visible clouding of the the fluid-filled space located in the front of the eye between the cornea and the iris) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
subjects
  Baseline | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  Day 14 | 0 | 0 | 0 | 0
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Day 90 | 0 | 0 | 0 | 0
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Day 180 | 0 | 0 | 0 | 0
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 0 | 0 | 0 | 0
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 0 | 0 | 0 | 0

51. Primary Outcome: Number of Subjects With Clinically Significant Biomicroscopy Findings as Determined by the Investigator at Each Study Visit - Lens Opacity
Description: An eye exam (slit lamp biomicroscopy) was performed by the investigator at each study visit. Findings related to lens opacity (a clouding of the eye's natural lens) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with natural lens intact (phakic) and data at visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 137 | 137 | 74 | 74
Number analyzed (eye) | 137 | 137 | 74 | 74
subjects
  Baseline | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 130 | 130 | 69 | 69
  Day 14: number analyzed (eye) | 130 | 130 | 69 | 69
  Day 14 | 0 | 0 | 0 | 0
  Day 90: number analyzed (Participants) | 125 | 126 | 66 | 66
  Day 90: number analyzed (eye) | 125 | 126 | 66 | 66
  Day 90 | 0 | 0 | 0 | 0
  Day 180: number analyzed (Participants) | 108 | 110 | 59 | 60
  Day 180: number analyzed (eye) | 108 | 110 | 59 | 60
  Day 180 | 0 | 0 | 0 | 0
  Day 270: number analyzed (Participants) | 105 | 105 | 57 | 57
  Day 270: number analyzed (eye) | 105 | 105 | 57 | 57
  Day 270 | 0 | 0 | 0 | 0
  Day 365: number analyzed (Participants) | 106 | 107 | 59 | 59
  Day 365: number analyzed (eye) | 106 | 107 | 59 | 59
  Day 365 | 0 | 0 | 0 | 0

52. Primary Outcome: Mean Total Ocular Staining Score by Visit
Description: Total corneal (fluorescein) staining score ranges between 0 and 5. Total conjunctival staining score is collected as the sum of lissamine green staining nasal and temporal scores and ranges between 0 and 10 per eye. Total ocular staining score is collected as the sum of total corneal and conjunctival scores (0 to 15) with a maximum possible score of 15 per eye. A higher total score indicates greater staining (or worse condition).
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
score on a scale
  Baseline | 4.08 (2.167) | 4.36 (2.332) | 3.77 (2.163) | 4.02 (2.352)
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  Day 14 | 3.46 (2.339) | 3.70 (2.395) | 3.45 (2.368) | 3.64 (2.400)
  Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Day 90 | 2.91 (2.415) | 3.17 (2.543) | 2.97 (2.674) | 3.27 (2.815)
  Day 180: number analyzed (Participants) | 153 | 153 | 75 | 75
  Day 180: number analyzed (eye) | 153 | 153 | 75 | 75
  Day 180 | 2.74 (2.493) | 2.85 (2.518) | 2.65 (2.477) | 3.05 (2.663)
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 2.45 (2.513) | 2.78 (2.556) | 2.53 (2.524) | 2.86 (2.516)
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 2.97 (2.841) | 2.97 (2.625) | 2.89 (2.619) | 3.30 (2.807)

53. Primary Outcome: Mean Intraocular Pressure by Visit
Description: Intraocular pressure was measured using Goldmann applanation tonometry and measured in millimeters mercury (mmHg). Values between 10mmHg and 20mmHg are considered normal eye pressure.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at visit
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 182 | 182 | 93 | 93
Number analyzed (eye) | 182 | 182 | 93 | 93
mmHg
  Baseline | 15.4 (2.48) | 15.6 (2.57) | 15.5 (2.75) | 15.6 (2.71)
  Day 14: number analyzed (Participants) | 175 | 175 | 88 | 88
  Day 14: number analyzed (eye) | 175 | 175 | 88 | 88
  Day 14 | 15.5 (2.82) | 15.6 (2.85) | 15.6 (2.81) | 15.5 (2.86)
  9Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  9Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  9Day 90 | 15.6 (2.52) | 15.5 (2.61) | 15.2 (2.72) | 15.0 (2.86)
  Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Day 180 | 15.5 (2.62) | 15.7 (2.62) | 14.8 (2.68) | 14.8 (2.66)
  Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Day 270 | 15.3 (2.66) | 15.5 (2.49) | 15.1 (2.79) | 15.2 (2.98)
  Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Day 365 | 15.4 (2.55) | 15.4 (2.77) | 15.4 (3.15) | 15.5 (3.06)

54. Primary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Dilated Fundus Exam Results by Visit - Vitreous
Description: An examination of the back of the eye (dilated fundus exam) was performed by the investigator. Findings related to the vitreous (the clear gel that fills the space between the lens and the retina of the eyeball) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 174 | 174 | 88 | 88
Number analyzed (eye) | 174 | 174 | 88 | 88
subjects
  Clinically Significant Change from Baseline at Day 14 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270 | 0 | 0 | 1 | 0
  Clinically Significant Change from Baseline at Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365 | 0 | 0 | 1 | 0

55. Primary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Dilated Fundus Exam Results by Visit - Retina
Description: An examination of the back of the eye (dilated fundus exam) was performed by the investigator. Findings related to the retina (the light-sensitive tissue lining the back of the eye that converts light into electrical signals the brain then interprets as images) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 174 | 174 | 88 | 88
Number analyzed (eye) | 174 | 174 | 88 | 88
subjects
  Clinically Significant Change from Baseline at Day 14 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365 | 0 | 0 | 0 | 1

56. Primary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Dilated Fundus Exam Results by Visit - Macula
Description: An examination of the back of the eye (dilated fundus exam) was performed by the investigator. Findings related to the macula (the round area at the center of the retina that provides central vision) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 174 | 174 | 88 | 88
Number analyzed (eye) | 174 | 174 | 88 | 88
subjects
  Clinically Significant Change from Baseline at Day 14 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270 | 0 | 0 | 1 | 0
  Clinically Significant Change from Baseline at Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365 | 0 | 0 | 1 | 0

57. Primary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Dilated Fundus Exam Results by Visit - Optic Nerve
Description: An examination of the back of the eye (dilated fundus exam) was performed by the investigator. Findings related to the optic nerve (the nerve that transmits visual information from the retina to the brain) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 174 | 174 | 88 | 88
Number analyzed (eye) | 174 | 174 | 88 | 88
subjects
  Clinically Significant Change from Baseline at Day 14 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365 | 0 | 0 | 0 | 0

58. Primary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Dilated Fundus Exam Results by Visit - Choroid
Description: An examination of the back of the eye (dilated fundus exam) was performed by the investigator. Findings related to the choroid (the layer of blood vessels and connective tissue between the white of the eye and retina) were graded as Normal or Abnormal. Abnormal findings were categorized as clinically significant (CS) or not clinically significant (NCS). CS findings were defined at those that may interfere with study parameters or otherwise confound the data as determined by the investigator.
Time Frame: Baseline (Day 1 pretreatment), Day 14, Day 90, Day 180, Day 270, Day 365
Population: Safety Population with data at baseline and corresponding visit
Measure: Number; unit: subjects
Units Other Than Participants: eye
Arm/Group | 0.003% AR-15512 - Right Eye | 0.003% AR-15512 - Left Eye | AR-15512 Vehicle - Right Eye | AR-15512 Vehicle - Left Eye
Number analyzed (Participants) | 174 | 174 | 88 | 88
Number analyzed (eye) | 174 | 174 | 88 | 88
subjects
  Clinically Significant Change from Baseline at Day 14 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 90: number analyzed (Participants) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90: number analyzed (eye) | 169 | 169 | 84 | 84
  Clinically Significant Change from Baseline at Day 90 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 180: number analyzed (Participants) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180: number analyzed (eye) | 153 | 153 | 76 | 76
  Clinically Significant Change from Baseline at Day 180 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 270: number analyzed (Participants) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270: number analyzed (eye) | 148 | 148 | 74 | 74
  Clinically Significant Change from Baseline at Day 270 | 0 | 0 | 0 | 0
  Clinically Significant Change from Baseline at Day 365: number analyzed (Participants) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365: number analyzed (eye) | 149 | 149 | 76 | 76
  Clinically Significant Change from Baseline at Day 365 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: An adverse event was (AE) defined as any untoward medical occurrence associated with the administration of the drug in humans, whether or not considered to be related to the study intervention. AEs were collected from time of consent until study exit, approximately 1 year. On the day of consent, randomized treatment was initiated.
Description: All participants were monitored for serious and other ocular and non-ocular AEs. All-Cause Mortality was not monitored for the ocular arms. However, the non-ocular AE arms were not considered at risk for ocular adverse event terms as the arms are reporting non-ocular-specific AEs. Similarly, the ocular AE arms were not considered at risk for non-ocular adverse event terms as the arms are reporting ocular-specific AEs.
Groups:
- 0.003% AR-15512 Ocular; 0.003% AR-15512 Non-ocular: 0.003% AR-15512 ophthalmic solution, one drop in each eye twice a day for 365 days
- AR-15512 Vehicle Ocular; AR-15512 Vehicle Non-ocular: AR-15512 vehicle ophthalmic solution, one drop in each eye twice a day for 365 days
Arm/Group | 0.003% AR-15512 Ocular | 0.003% AR-15512 Non-ocular | AR-15512 Vehicle Ocular | AR-15512 Vehicle Non-ocular
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/182 | 0/0 | 0/93
Serious Adverse Events (participants affected / at risk) | 1/182 | 6/182 | 2/93 | 6/93
Other Adverse Events (participants affected / at risk) | 90/182 | 0/182 | 7/93 | 0/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 0.003% AR-15512 Ocular (N=182) | 0.003% AR-15512 Non-ocular (N=182) | AR-15512 Vehicle Ocular (N=93) | AR-15512 Vehicle Non-ocular (N=93)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 0/0 | 1 (1) | 0/0
Retinal detachment (Eye disorders) | 0 (0) | 0/0 | 1 (1) | 0/0
Retinal tear (Eye disorders) | 1 (1) | 0/0 | 0 (0) | 0/0
Small intestinal obstruction (Gastrointestinal disorders) | 0/0 | 0 (0) | 0/0 | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0/0 | 1 (1) | 0/0 | 0 (0)
Cellulitis (Infections and infestations) | 0/0 | 0 (0) | 0/0 | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0/0 | 0 (0) | 0/0 | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0/0 | 1 (1) | 0/0 | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0/0 | 0 (0) | 0/0 | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0/0 | 0 (0) | 0/0 | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0/0 | 0 (0) | 0/0 | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 1 (1) | 0/0 | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 1 (1) | 0/0 | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 1 (1) | 0/0 | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0/0 | 1 (1) | 0/0 | 0 (0)
Syncope (Nervous system disorders) | 0/0 | 0 (0) | 0/0 | 1 (1)
Hypotension (Vascular disorders) | 0/0 | 1 (1) | 0/0 | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 0.003% AR-15512 Ocular (N=182) | 0.003% AR-15512 Non-ocular (N=182) | AR-15512 Vehicle Ocular (N=93) | AR-15512 Vehicle Non-ocular (N=93)
Instillation site pain (General disorders) | 90 | 0/0 | 7 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT05493111/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT05493111/SAP_001.pdf